CLINICAL TRIAL: NCT02280980
Title: Effectiveness of Oculomotor and Gaze Stability Exercises on the Improvement of Balance After Brain Stroke in Patients Older Than 60 Years Old
Brief Title: Effect of Oculomotor and Gaze Stability Exercises on the Improvement of Balance After Stroke
Acronym: BETTERBALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLC.CI.HCC7.2014
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Distorted; Balance
Keywords: Stroke; Postural Balance; Oculomotor and Gaze Stability Exercises; Rehabilitation; Physical therapy; Outpatient
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined rehabilitation protocol (Experimental): The usual rehabilitation protocol in the physiotherapy department is supplemented with a three weeks home protocol of oculomotor and gaze stability exercises.
  Interventions: Other: Oculomotor and Gaze Stability Exercises
- Usual rehabilitation protocol (No Intervention): The usual rehabilitation protocol in the physiotherapy department for patients after stroke.

INTERVENTIONS:
Other: Oculomotor and Gaze Stability Exercises — Daily oculomotor and gaze stability exercises, twice a day, for three weeks
  Arms: Combined rehabilitation protocol

SUMMARY:
Individuals older than 60 years old, discharged after suffering brain stroke with referral to the rehabilitation outpatient clinic, will be assessed for orthostatic balance. Patients with positive Romberg test are invited to participate in the trial. Participants will be randomized to either the current rehabilitation protocol or to an supplemental intervention focused on oculomotor and gaze stability exercises to be applied at home for three weeks. Participants will be assessed with standardized, validated tools.

DETAILED DESCRIPTION:
The study aims to evaluated the effect of a home program of oculomotor and gaze stability exercises on improvement the balance in stroke patients.

Individuals older than 60 years old, discharged after suffering brain stroke and referred to the neurologic rehabilitation outpatient clinic, will be assessed for a neuro-motor deficits. Patients will be consider eligible if they had positive Romberg test (disorder of orthostatic balance) and they will be invited to participate in the trial. Patients with previous balance problems will be excluded.

Participants will be allocated in two intervention groups through block randomization, either the current rehabilitation protocol or to an supplemental intervention focused on oculomotor and gaze stability exercises to be applied at home for three weeks. Participants will be assessed with Motor Assessment Scale, Berg Balance Scale and Timed Up and Go Test.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis 3 to 15 months before recruitment
* Balance deficits (positive Romberg)
* Patients able to walk 3 meters without assistance with or without an assistive device

Exclusion Criteria:

* Balance problems previous to the index stroke
* Severe osteo-articular lesions that compromise the ability to perform the proposed exercises
* Previous exposure to oculomotor or gaze stability exercises

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Change on BBS from baseline up to three weeks of intervention
  Balance measure used in older people with impairment in balance function by assessing the performance of functional tasks
Timed Up and Go Test (TUG) | Change on TUG from baseline up to three weeks of intervention
  simple test used to assess mobility and requires both static and dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Correia, Pt, MSc, Principal Investigator — Centro Hospitalar de Lisboa Central; Carla Pimenta, Pt, MSc, Principal Investigator — Centro Hospitalar de Lisboa Central

IPD SHARING:
Plan to Share IPD: Yes
Patients are informed that their records are available to them.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Berg, K., Wood-Dauphinée, S., Williams, J. & Gayton, D. (1989). Measuring balance in the elderly: preliminary development of an instrument. Physiotherapy Canada, 41, 304-311.
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Carr JH, Shepherd RB, Nordholm L, Lynne D. Investigation of a new motor assessment scale for stroke patients. Phys Ther. 1985 Feb;65(2):175-80. doi: 10.1093/ptj/65.2.175. PMID 3969398
- [Background] Dias et al (2009). Aplicação da Escala de Equilíbrio de Berg para verificação do equilíbrio de idosos em diferentes fases do envelhecimento. RBCEH, 6(2), 213-224.
- [Background] Geurts AC, de Haart M, van Nes IJ, Duysens J. A review of standing balance recovery from stroke. Gait Posture. 2005 Nov;22(3):267-81. doi: 10.1016/j.gaitpost.2004.10.002. Epub 2004 Dec 7. PMID 16214666
- [Background] Hiengkaew V, Jitaree K, Chaiyawat P. Minimal detectable changes of the Berg Balance Scale, Fugl-Meyer Assessment Scale, Timed "Up & Go" Test, gait speeds, and 2-minute walk test in individuals with chronic stroke with different degrees of ankle plantarflexor tone. Arch Phys Med Rehabil. 2012 Jul;93(7):1201-8. doi: 10.1016/j.apmr.2012.01.014. Epub 2012 Apr 12. PMID 22502805
- [Background] Morimoto H, Asai Y, Johnson EG, Lohman EB, Khoo K, Mizutani Y, Mizutani T. Effect of oculo-motor and gaze stability exercises on postural stability and dynamic visual acuity in healthy young adults. Gait Posture. 2011 Apr;33(4):600-3. doi: 10.1016/j.gaitpost.2011.01.016. Epub 2011 Feb 19. PMID 21334899
- [Derived] Correia A, Pimenta C, Alves M, Virella D. Better balance: a randomised controlled trial of oculomotor and gaze stability exercises to reduce risk of falling after stroke. Clin Rehabil. 2021 Feb;35(2):213-221. doi: 10.1177/0269215520956338. Epub 2020 Sep 9. PMID 32907392
- [Derived] Pimenta C, Correia A, Alves M, Virella D. Effects of oculomotor and gaze stability exercises on balance after stroke: Clinical trial protocol. Porto Biomed J. 2017 May-Jun;2(3):76-80. doi: 10.1016/j.pbj.2017.01.003. Epub 2017 Feb 12. PMID 32258591